CLINICAL TRIAL: NCT05456828
Title: A Multi-Center, Open-label, Single Ascending-Dose and Multiple Ascending-Dose Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ASKG712 Following Intravitreal Administration in Patients With Neovascular Age-related Macular Degeneration
Brief Title: A Study of ASKG712 in Patients With Neovascular Age-Related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AskGene Pharma, Inc. (Industry)
Collaborators: Suzhou Aosaikang Biopharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASKG712-CT-I-1
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASKG712 (Experimental): Single or multiple ascending dose of ASKG712 by intravitreal injection
  Interventions: Biological: ASKG712

INTERVENTIONS:
Biological: ASKG712 — ASKG712 is a recombinant anti-VEGF humanized monoclonal antibody and Ang-2 antagonist peptide fusion protein, which has high specificity for the binding of VEGF-A and Ang-2.
  Other Names: AM712

SUMMARY:
The purpose of the Phase 1 study is comprised of single ascending-dose component (Part 1) , multiple ascending-dose component (Part 2) and multiple-dose extension component (Part 3) to evaluate the safety, tolerability, pharmacokinetics, and efficacy of ASKG712 in patients with neovascular age-related macular degeneration (nAMD).

DETAILED DESCRIPTION:
The Part 1 of study is a multicenter, open-label, sequentially, single ascending-dose study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of ASKG712 in subjects with nAMD.

The Part 2 of study is a multicenter, open-label, sequentially, multiple ascending-dose (3 doses) study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of ASKG712 in subjects with nAMD.

The Part 3 of study is a multicenter, open-label, randomized, multiple ascending-dose (3 doses) study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of ASKG712 in subjects with nAMD at 2 recommanded dose levels.

Subjects will be sequentially enrolled into different dose-level cohorts following the "3+3" design to determine the maximum tolerated dose (MTD) or the maximum administered dose has been reached.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed the informed consent form;
* 2. Male or female subjects with 50~80 years of age;
* 3. Active sub-foveal or juxta-foveal choroidal neovascularization(CNV) lesions secondary to neovascular age-related macular degeneration(nAMD);
* 4. Total lesion area ≤ 12 disc area(DA);
* 5. BCVA letter score measured at screening of 19~78 letters.

Exclusion Criteria:

* 1. History of uveitis in either eye；
* 2. Current active inflammation or infection in the study eye;
* 3. Central foveal scar, fibrosis or atrophy of macular in the study eye;
* 4. Subretinal hemorrhage area in the study eye ≥ 50% of total lesion size;
* 5. Scar or fibrosis area in study eyes ≥ 50% of total lesion size;
* 6. History or any concurrent ocular condition which, in opinion of investigator, could either confound interpretation of efficacy and safety of ASKG712 or require medical or surgical intervention.
* 7. Presence of retinal pigment epithelial tear;
* 8. Previous intraocular operations in the study eye;
* 9. Uncontrolled previous or current glaucoma in either eye, or previous glaucoma filtering operation in the study eye;
* 10. Previous anti-VEGF drug treatment within 60 days prior to screening；
* 11. Diseases that affect intravenous injection and venous blood sampling;
* 12. Systemic autoimmune diseases;
* 13. Any uncontrolled clinical disorders;
* 14. History of allergy or current allergic response to ASKG712 or fluorescein;
* 15. Pregnant or nursing women;
* 16. Subjects should be excluded in the opinion of investigators.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular adverse events (AEs) of the study eyes | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: up to 36 weeks
  Any relevant ocular observations assessed by best corrected visual acuity (BCVA) , slitlamp examination, ophthalmoscopy, intraocular pressure, fundus photography, optical coherence tomography (OCT) and angiography
Incidence of non-ocular adverse events (AEs) | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: up to 36 weeks
  Any changes of clinical safety observations assessed by vital signs, electrocardiograph (ECG), clinical laboratory tests and physical examination

SECONDARY OUTCOMES:
Area under the concentration time curve (AUC) | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: 20 weeks
  To evaluate the systemic pharmacokinetics of ASKG712 in subjects with neovascular age-related macular degenerationn (nAMD)
Maximum plasma concentration (Cmax) | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: 20 weeks
  To evaluate the systemic pharmacokinetics of ASKG712 in subjects with neovascular age-related macular degenerationn (nAMD)
Anti-Drug Antibody | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: 20 weeks
  To evaluate the immunogenicity of ASKG712 in subjects with neovascular age-related macular degenerationn (nAMD)
Mean change from baseline in best corrected visual acuity (BCVA) as measured by Early Treatment of Diabetic Retinopathy Study (ETDRS) letter score | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: up to 36 weeks
  To evaluate the efficacy of ASKG712 in subjects with neovascular age-related macular degenerationn (nAMD)
Mean change from baseline in central subfield thickness (CST) of macula measured by optical coherence tomography (OCT) | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: up to 36 weeks
  To evaluate the efficacy of ASKG712 in subjects with neovascular age-related macular degenerationn (nAMD)
Mean change from baseline in choroidal neovascularization area measured by fundus angiography | Part 1: 6 weeks; Part 2: 20 weeks; Part 3: 20 weeks
  To evaluate the efficacy of ASKG712 in subjects with neovascular age-related macular degenerationn (nAMD)

CONTACTS AND LOCATIONS:
Overall Officials: Kun Liu, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD or supporting information available.